CLINICAL TRIAL: NCT02260934
Title: Rituximab Plus Cyclophosphamide Followed by Belimumab for the Treatment of Lupus Nephritis (ITN055AI)
Brief Title: Rituximab and Belimumab for Lupus Nephritis
Acronym: CALIBRATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN055AI; CALIBRATE (Other: Immune Tolerance Network)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Rituximab; Cyclophosphamide; Prednisone; Methylprednisolone; Methylprednisolone Hemisuccinate; Diphenhydramine; Acetaminophen; belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab/Cyclophosphamide (RC) (Active Comparator): Prednisone taper to 10 mg/day by week 12 and continue prednisone 10 mg/day to week 96.
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Methylprednisolone; Drug: Diphenhydramine; Drug: Acetaminophen
- Rituximab/Cyclophosphamide/Belimumab (RCB) (Experimental): 1. Belimumab (10 mg/kg IV) at weeks 4, 6, 8, and every 4 weeks to week 48.
  2. Prednisone taper to 10 mg/day by week 12, and continue prednisone 10 mg/day to week 96.
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Methylprednisolone; Drug: Diphenhydramine; Drug: Acetaminophen; Biological: Belimumab

INTERVENTIONS:
Biological: Rituximab — Rituximab 1000mg intravenously (IV) at week 0 and week 2
  Other Names: Rituxan
  Arms: Rituximab/Cyclophosphamide (RC)
Drug: Cyclophosphamide — Cyclophosphamide (750 mg) intravenously (IV) at week 0 and week 2.
  Other Names: Cytoxan
  Arms: Rituximab/Cyclophosphamide (RC)
Drug: Prednisone — * Week 0 and Week 2: Prednisone (40 mg/day; taper to 10 mg/day by week 12)
  * Continue prednisone 10 mg/day to week 96
  Other Names: Deltasone
  Arms: Rituximab/Cyclophosphamide (RC)
Drug: Methylprednisolone — Week 0 and Week 2:
  Solumedrol (100 mg) IV
  Other Names: Solu-Medrol
  Arms: Rituximab/Cyclophosphamide (RC)
Drug: Diphenhydramine — Diphenhydramine (50 mg, or equivalent dose of similar antihistamine) will be given orally 1 hour (plus or minus 15 minutes) before each infusion of rituximab.
  Arms: Rituximab/Cyclophosphamide (RC)
Drug: Acetaminophen — Acetaminophen (650 mg) will be given orally 1 hour (plus or minus 15 minutes) before each infusion of rituximab.
  Other Names: Tylenol
  Arms: Rituximab/Cyclophosphamide (RC)
Biological: Rituximab — Rituximab 1000mg intravenously (IV) at week 0 and week 2.
  Other Names: Rituxan
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)
Drug: Cyclophosphamide — Cyclophosphamide (750 mg) intravenously (IV) at week 0 and week 2.
  Other Names: Cytoxan
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)
Drug: Prednisone — * Week 0 and Week 2: Prednisone (40 mg/day; taper to 10 mg/day by week 12)
  * Continue prednisone 10 mg/day to week 96
  Other Names: Deltasone
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)
Drug: Methylprednisolone — Week 0 and Week 2: Solumedrol (100 mg) IV
  Other Names: Solu-Medrol
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)
Drug: Diphenhydramine — Diphenhydramine (50 mg, or equivalent dose of similar antihistamine) will be given orally 1 hour (plus or minus 15 minutes) before each infusion of rituximab.
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)
Drug: Acetaminophen — Acetaminophen (650 mg) will be given orally 1 hour (plus or minus 15 minutes) before each infusion of rituximab.
  Other Names: Tylenol
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)
Biological: Belimumab — The RCB Group will receive IV belimumab 10mg/kg at weeks 4, 6, 8, and then every 4 weeks through week 48
  Other Names: Benlysta
  Arms: Rituximab/Cyclophosphamide/Belimumab (RCB)

SUMMARY:
In this experimental study, researchers will try to find out if treatment of lupus nephritis with a combination of rituximab and cyclophosphamide (CTX), or a combination of rituximab and CTX followed by treatment with belimumab is safe and if this drug combination can block the immune system attacks.

DETAILED DESCRIPTION:
Lupus nephritis is a severe form of systemic lupus erythematosus (SLE) with active disease in the kidneys. SLE is a complex disease in which the body's own immune system attacks some of the body parts: the skin, the joints, the kidneys, the nervous system, the heart, the lungs and the blood. The cause of SLE is not known. Treatment for SLE usually involves drugs that are designed to block the immune system attacks. When SLE affects the kidneys (nephritis), stronger immune suppressing treatment is usually needed.

The drugs used in treatment of lupus nephritis often do not cure the disease and can cause serious side effects, including lowering the immune system too much. When the immune system is too low, a person is at a higher risk of getting infections. Therefore, research into new treatments with fewer serious side effects is needed for lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Systemic Lupus Erythematosus (SLE) by American College of Rheumatology (ACR) criteria.
2. Positive antinuclear antibody (ANA) or positive anti-ds DNA test results at visit -1 or any time within 14 days before visit -1.
3. Active proliferative lupus nephritis, as defined by either of the following:

   * Kidney biopsy documentation within the last 3 months of International Society of Nephrology/Renal Pathology Society (ISN/RPS) proliferative nephritis: Class III, Class IV, or Class V in combination with Class III or IV.
   * Active urinary sediment and kidney biopsy documentation within the last 12 months of ISN/RPS proliferative nephritis: Class III, Class IV, or Class V in combination with Class III or IV. Active urinary sediment is defined as any one of the following:
   * >5 RBC/hpf in the absence of menses and infection;
   * >5 White blood cell per high powered field (WBC/hpf) in the absence of infection; or
   * Cellular casts limited to RBC or WBC casts.
4. Urine protein-to-creatinine ratio (UPCR) >1 at study entry based on a 24-hour collection.
5. Ability to provide informed consent.

Exclusion Criteria:

1. New onset lupus nephritis, defined as lupus nephritis for which the participant has not yet been treated with either mycophenolate mofetil or cyclophosphamide.
2. Neutropenia (absolute neutrophil count <1500/mm^3).
3. Thrombocytopenia (platelets <50,000/mm^3).
4. Moderately severe anemia (Hgb < mg/dL).
5. Moderately severe hypogammaglobulinemia (IgG <450 mg/dL) or Immunoglobulin A (IgA) <10mg/dL.
6. Positive QuantiFERON -Tuberculosis (TB) Gold test results.
7. Pulmonary fibrotic changes on chest radiograph consistent with prior healed tuberculosis.
8. Active bacterial, viral, fungal, or opportunistic infections.
9. Evidence of infection with human immunodeficiency virus (HIV), hepatitis B (as assessed by HBsAg and anti-HBc) or hepatitis C.
10. Hospitalization for treatment of infections, or parenteral (IV or IM) antibacterials, antivirals, anti-fungals, or anti-parasitic agents within the past 60 days.
11. Chronic infection that is currently being treated with suppressive antibiotic therapy, including but not limited to tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria.
12. History of significant infection or recurrent infection that, in the investigator's opinion, places the participant at risk by participating in this study.
13. Receipt of a live-attenuated vaccine within 3 months of study enrollment.
14. End-stage renal disease (eGFR <20 mL/min/1.73m^2).
15. Concomitant malignancies or a history of malignancy, with the exception of adequately treated basal and squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
16. History of transplantation.
17. History of primary immunodeficiency.
18. Pregnancy.
19. Breastfeeding.
20. Unwillingness to use an FDA-approved form of birth control (including but not limited to a diaphragm, an intrauterine device, progesterone implants or injections, oral contraceptives, the double-barrier method, or a condom).
21. Use of cyclophosphamide within the past 6 months.
22. Use of anti-Tumor Necrosis Factor (TNF) medication, other biologic medications, or experimental non- biologic therapeutic agents within the past 90 days, or 5 half-lives prior to screening, whichever is greater.
23. Intravenous immunoglobulin (IVIG), plasmapheresis, or leukopheresis within the past 90 days.
24. Use of investigational biologic agent within the past 12 months.
25. Prior treatment with rituximab, belimumab, atacicept, or other biologic B cell therapy.
26. Liver function test [aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase] results that are >=2 times the upper limit of normal.
27. Severe, progressive, or uncontrolled renal, hepatic, hematological,gastrointestinal, pulmonary, cardiac, or neurological disease, either related or unrelated to SLE, with the exception of active lupus nephritis (or, in the investigator's opinion, any other concomitant medical condition that places the participant at risk by participating in this study).
28. Comorbidities requiring corticosteroid therapy, including those which have required three or more courses of systemic corticosteroids within the previous 12 months.
29. Current substance abuse or history of substance abuse within the past year.
30. History of severe allergic or anaphylactic reactions to chimeric or fully human monoclonal antibodies.
31. History of anaphylactic reaction to parenteral administration of contrast agents.
32. Lack of peripheral venous access.
33. History of severe depression or severe psychiatric condition.
34. History of suicidal thoughts within the past 2 months or suicidal behavior within the past 6 months, or a significant suicide risk in the investigator's opinion.
35. Inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Diamond, M.D., Study Chair — Feinstein Institute for Medical Research; David Wofsy, M.D., Study Chair — University of California San Francisco, Department of Medicine; Maria Dall'Era, M.D., Study Chair — University of California San Francisco, Department of Medicine; Cynthia Aranow, M.D., Study Chair — Feinstein Institute for Medical Research
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver: School of Medicine: Division of Rheumatology, Aurora, Colorado
  - Colorado Kidney Care, Denver, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Washington University in St. Louis, St Louis, Missouri
  - Feinstein Institute, North Shore Hospital, Manhasset, New York
  - New York University, Langone Medical Center, New York, New York
  - Weill Cornell Medical College: Hospital for Special Surgery -, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina School of Medicine:, Chapel Hill, North Carolina
  - Ohio State University Wexner Medical Center:, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access will be made available to the public at some point in the future via the mechanisms of : 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal.
Time Frame: The aim is to share IPD within 24 months upon study completion.
Access Criteria: ImmPort public data access.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- [Result] Atisha-Fregoso Y, Malkiel S, Harris KM, Byron M, Ding L, Kanaparthi S, Barry WT, Gao W, Ryker K, Tosta P, Askanase AD, Boackle SA, Chatham WW, Kamen DL, Karp DR, Kirou KA, Sam Lim S, Marder B, McMahon M, Parikh SV, Pendergraft WF 3rd, Podoll AS, Saxena A, Wofsy D, Diamond B, Smilek DE, Aranow C, Dall'Era M. Phase II Randomized Trial of Rituximab Plus Cyclophosphamide Followed by Belimumab for the Treatment of Lupus Nephritis. Arthritis Rheumatol. 2021 Jan;73(1):121-131. doi: 10.1002/art.41466. Epub 2020 Dec 1. PMID 32755035
- See also: National Institute of Allergy and Infectious Diseases website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org/
- See also: ITN CALIBRATE study website — http://calibratestudy.org/about-calibrate

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 59 participants screened, 43 were enrolled at 14 sites in the US from July 9, 2015 to May 22, 2017.
Pre-assignment Details: Prior to randomization, enrolled participants received infusions of Solumedrol 100mg, rituximab 1000mg, and cyclophosphamide 750mg intravenously (IV) at Week 0 and Week 2. Prednisone was administered at 40 mg/day for the first 2 weeks, followed by a guided steroid taper. Participants were randomized at Week 4.
Groups:
- Rituximab/Cyclophosphamide (RC): Participants received infusions of Solumedrol 100mg, rituximab 1000mg, and cyclophosphamide 750mg intravenously (IV) at Week 0 and Week 2. Prednisone was administered at 40 mg/day for the first 2 weeks, followed by a guided steroid taper to 10 mg/day by Week 12. Prednisone was continued through to Week 96 at 10 mg/day, with the potential of a taper to a minimum of 5 mg/day.
- Rituximab/Cyclophosphamide/Belimumab (RCB): Participants received infusions of Solumedrol 100mg, rituximab 1000mg, and cyclophosphamide 750mg intravenously (IV) at Week 0 and Week 2. Prednisone was administered at 40 mg/day for the first 2 weeks, followed by a guided steroid taper to 10 mg/day by Week 12. Prednisone was continued through to Week 96 at 10 mg/day, with the potential of a taper to a minimum of 5 mg/day. In addition, participants received IV belimumab 10mg/kg at Weeks 4, 6, 8, and then every 4 weeks through Week 48 in addition to prednisone.
Period: Overall Study
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Started | 22 | 21
Completed | 19 (At primary outcome timepoint: Ten participants engaged in ongoing scheduled study visits.) | 17 (At primary outcome timepoint: Eleven participants engaged in ongoing scheduled study visits.)
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Participant Relocated | 1 | 0
Not completed — Site error | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who signed informed consent and were enrolled in the study. Reported baseline measurements are the most recent measurements for a participant taken between the Screening Visit (occurring within 21 days of Week 0/Study Enrollment) and Week 0 (Study Enrollment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB) | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (11.4) | 34.5 (9.1) | 33.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 12 | 16 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 7 | 9 | 16
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 21 | 43
Urine Protein-to-Creatinine Ratio (UPCR) from 24 Hour Collection [Mean (Standard Deviation); unit: Ratio] — Urine protein-to-creatinine ratio (UPCR) from a 24-hour collection is a measure of lupus nephritis disease activity. Higher ratios indicate poorer kidney function. Elevated ratio: >3.
  Ratio | 3.4 (1.5) | 3.3 (2.5) | 3.4 (2.0)
Elevated Urine Protein-to-Creatinine Ratio (UPCR) [Count of Participants; unit: Participants] — Count of participants with a urine protein-to-creatinine ratio (UPCR) from a 24-hour collection that was >3.
  Participants | 14 | 8 | 22
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — Serum creatinine is a measure of renal function. Normal values: 0.67 to 1.18mg/dL for men and 0.51 to 0.95mg/dL for women. Higher results indicate poorer kidney function.
  mg/dL | 1.0 (0.4) | 1.0 (0.5) | 1.0 (0.4)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Estimated glomerular filtration rate (eGFR) is a measure of renal function. Methodology: Calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula based on serum creatinine, age, sex and race. Normal GFR: ≥90 mL/min/1.73m^2. Lower GFRs reflect poorer kidney function.
  mL/min/1.73m^2 | 92.7 (36.0) | 89.1 (33.9) | 90.9 (34.6)
Serum Albumin [Mean (Standard Deviation); unit: g/dL] — Normal values: 3.7 to 4.9 g/dL.
  g/dL | 3.0 (0.5) | 2.9 (0.6) | 2.9 (0.6)
B Cell Count [Mean (Standard Deviation); unit: cells/µL] — Total B cell number in the peripheral blood. B cell depletion was expected to occur in this study between Weeks 0 and 4, after initiation of rituximab and cyclophosphamide. Normal B Cell Count in the peripheral blood: 107 to 698 cells/µL. Population: Participants who signed informed consent and were enrolled in the study. Reported baseline measurements are the most recent measurements for a participant taken between the screening visit and Week 0.
  cells/µL
    number analyzed (Participants) | 18 | 18 | 36
    (all) | 160.5 (157.4) | 216.0 (207.3) | 188.3 (183.6)
Immunoglobulin G (IgG) Level [Mean (Standard Deviation); unit: mg/dL] — Immunoglobulin G (IgG) is a measure of immune function. Normal values: 700 to 1600 mg/dL.
  mg/dL | 1044.9 (408.9) | 1057.1 (589.5) | 1050.8 (499.1)
Hypogammaglobulinemia [Count of Participants; unit: Participants] — Count of participants with hypogammaglobulinemia at baseline, defined as having a serum Immunoglobulin G (IgG) level <450 mg/dL.
  Participants | 2 | 4 | 6
Anti-Double Stranded DNA (Anti-dsDNA) Positive [Count of Participants; unit: Participants] — Count of participants who were anti-double stranded DNA (anti-dsDNA) positive at baseline, defined as anti-dsDNA levels >30 IU/mL. Anti-dsDNA levels are associated with systemic lupus erythematosus disease activity.
  Participants | 20 | 19 | 39
Hypocomplementemic for C3 [Count of Participants; unit: Participants] — Count of participants who were hypocomplementemic for C3, defined as a C3 level <90 mg/dL. Serum C3 complement is a protein which can be measured in the blood. Low blood levels of C3 are common in those with active lupus.
  Participants | 18 | 16 | 34
Hypocomplementemic for C4 [Count of Participants; unit: Participants] — Count of participants who were hypocomplementemic for C4, defined as C4 level <10 mg/dL. Serum C4 complement is a protein which can be measured in the blood. Low blood levels of C4 are common in those with active lupus.
  Participants | 10 | 8 | 18
Weight [Mean (Standard Deviation); unit: kg] — Body weight measurement taken before infusion of study drug.
  kg | 69.7 (18.0) | 75.4 (26.0) | 72.5 (22.2)
Duration of Lupus Nephritis [Mean (Standard Deviation); unit: Years] — Duration of lupus nephritis (LN) is the number of years at the screening visit since the onset of LN.
  Years | 4.8 (4.5) | 6.8 (6.6) | 5.8 (5.7)
Duration of Lupus Nephritis More Than One Year [Count of Participants; unit: Participants] — Count of participants with a duration of lupus nephritis of greater than one year. Duration of lupus nephritis is defined by the number of years from onset of lupus nephritis to the screening visit.
  Participants
    > 1 year | 18 | 18 | 36
    ≤ 1 year | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Grade 3 or Higher Infectious Adverse Event By Week 24, Week 48 and Week 96
Description: The percentage of participants who experienced at least one Grade 3 or higher treatment-emergent infectious adverse event. The severity of adverse events (AEs) was classified into grades using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, v4.03:June 14, 2010). Treatment-emergent AEs are those:
  * with an onset date on or after the first dose of study medication,
  * with onset before first dose but that worsened in severity after first dose, and
  * for which the start of the AE in relation to the start of study medication could not be established.
  AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 17.0. Grade 3 or higher AEs were classified infectious based on the study team's review of the MedDRA body systems and preferred terms of the AEs.
Time Frame: Week 0 to Week 96
Population: The modified intent-to-treat population includes all randomized participants who received 1 dose of Solumedrol, 1 dose of rituximab, 1 dose of cyclophosphamide, and, if in the Rituximab/Cyclophosphamide/Belimumab (RCB) arm, 1 dose of belimumab.
  Confidence intervals were calculated using Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 0 to Week 24 | 9.1 [1.1 to 29.2] | 4.8 [0.1 to 23.8]
  Week 0 to Week 48 | 22.7 [7.8 to 45.4] | 9.5 [1.2 to 30.4]
  Week 0 to Week 96 | 27.3 [10.7 to 50.2] | 9.5 [1.2 to 30.4]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 24; Test type: Superiority; p = 0.58, Regression, Logistic — Two-sided test; Treatment group was the independent variable in the logistic regression
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 48; Test type: Superiority; p = 0.25, Regression, Logistic — Two-sided test; Treatment group was the independent variable in the logistic regression
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 96; Test type: Superiority; p = 0.15, Regression, Logistic — Two-sided test; Treatment group was the independent variable in the logistic regression

2. Secondary Outcome: Percentage of Participants With B Cell Reconstitution at Week 24, Week 48 and Week 96
Description: The percentage of participants who achieved B cell reconstitution, defined as a peripheral blood total B cell count ≥ to the baseline count or the lower limit of normal, whichever was lower. Note: B cell depletion was expected to occur in this study between Weeks 0 and 4, after initiation of rituximab and cyclophosphamide.
  Normal peripheral blood B Cell count: 107 to 698 cells/µL.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
Percentage of Participants
  Week 24: number analyzed (Participants) | 16 | 16
  Week 24 | 31.3 [11.0 to 58.7] | 6.3 [0.2 to 30.2]
  Week 48: number analyzed (Participants) | 14 | 17
  Week 48 | 35.7 [12.8 to 64.9] | 11.8 [1.5 to 36.4]
  Week 96: number analyzed (Participants) | 15 | 13
  Week 96 | 40.0 [16.3 to 67.7] | 30.8 [9.1 to 61.4]

3. Secondary Outcome: Percentage of Participants With Grade 4 Hypogammaglobulinemia by Week 24, Week 48, and Week 96
Description: The percentage of participants who experienced Grade 4 hypogammaglobulinemia, defined as having a serum Immunoglobulin G (IgG) level < 300 mg/dL. Severity of adverse events (AEs) was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, v4.03:June 14, 2010).
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rituximab/Cyclophosphamide/Belimumab (RCB): Participants received infusions of Solumedrol 100mg, rituximab 1000mg, and cyclophosphamide 750mg intravenously (IV) at Week 0 and Week 2. Prednisone was administered at 40 mg/day for the first 2 weeks, followed by a guided steroid taper to 10 mg/day by Week 12. Prednisone was continued through to Week 96 at 10 mg/day, with the potential of a taper to a minimum of 5 mg/day.
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 0 to Week 24 | 0 [0.0 to 15.4] | 0 [0.0 to 16.1]
  Week 0 to Week 48 | 0 [0.0 to 15.4] | 0 [0.0 to 16.1]
  Week 0 to Week 96 | 0 [0.0 to 15.4] | 0 [0.0 to 16.1]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 24; Test type: Superiority — P-value could not be produced because of zero count in at least one of the treatment arms; Regression, Logistic; Two sided test. P-value could not be produced because of zero count in at least one of the treatment arms; Treatment group was the independent variable in the logistic regression
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 48; Test type: Superiority; Regression, Logistic; P-value could not be produced because of zero count in at least one of the treatment arms; P-value could not be produced because of zero count in at least one of the treatment arms
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 96 The modified intent to treat population includes all randomized participants who received 1 dose of Solumedrol, 1 dose of rituximab, 1 dose of cyclophosphamide, and, if in the Rituximab/Cyclophosphamide/Belimumab (RCB) arm, 1 dose of belimumab; Test type: Superiority — P-value could not be produced because of zero count in at least one of the treatment arms; Regression, Logistic; P-value could not be produced because of zero count in at least one of the treatment arms; P-value could not be produced because of zero count in at least one of the treatment arms

4. Secondary Outcome: Percentage of Participants With a Complete Response at Week 24, Week 48, and Week 96
Description: The percentage of participants who achieved a complete response, defined as meeting all of the following criteria:
  1. Urine protein-to-creatinine ratio (UPCR) < 0.5, based on a 24-hour collection;
  2. Estimated glomerular filtration rate (eGFR) ≥ 120 ml/min/1.73 m^2 calculated by the CKD-EPI formula or, if < 120 ml/min/1.73 m^2, then > 80% of eGFR at entry; and
  3. Prednisone dose tapered to 10 mg/day and adherence to prednisone dosing provisions.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rituximab/Cyclophosphamide (RC); Rituximab/Cyclophosphamide/Belimumab (RCB): The modified intent to treat population includes all randomized participants who received 1 dose of Solumedrol, 1 dose of rituximab, 1 dose of cyclophosphamide, and, if in the Rituximab/Cyclophosphamide/Belimumab (RCB) arm, 1 dose of belimumab.
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 24: number analyzed (Participants) | 21 | 20
  Week 24 | 23.8 [8.2 to 47.2] | 30.0 [11.9 to 54.3]
  Week 48: number analyzed (Participants) | 20 | 19
  Week 48 | 35.0 [15.4 to 59.2] | 42.1 [20.3 to 66.5]
  Week 96: number analyzed (Participants) | 15 | 14
  Week 96 | 33.3 [11.8 to 61.6] | 42.9 [17.7 to 71.1]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 24; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.66, Regression, Logistic — Treatment group was the independent variable in the logistic regression; 2 sided test
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 48; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.65, Regression, Logistic — Treatment group was the independent variable in the logistic regression; 2 sided test; Treatment group was the independent variable in the logistic regression

5. Secondary Outcome: Percentage of Participants With an Overall Response at Week 24, Week 48, and Week 96
Description: The percentage of participants who achieved an overall response, defined as meeting all of the following criteria:
  1. >50% improvement in the urine protein-to-creatinine ratio (UPCR) from study entry, based on a 24-hour collection;
  2. Estimated glomerular filtration rate (eGFR) ≥120 ml/min/1.73 m^2 calculated by the CKD-EPI formula or, if < 120 ml/min/1.73 m^2, then > 80% of eGFR at entry; and
  3. Prednisone dose tapered to 10 mg/day and adherence to prednisone dosing provisions.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 24: number analyzed (Participants) | 21 | 20
  Week 24 | 46.7 [25.7 to 70.2] | 55.0 [31.5 to 76.9]
  Week 48: number analyzed (Participants) | 20 | 19
  Week 48 | 60.0 [36.1 to 80.9] | 73.7 [48.8 to 90.9]
  Week 96: number analyzed (Participants) | 15 | 14
  Week 96 | 53.3 [26.6 to 78.7] | 71.4 [41.9 to 91.6]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 24 Treatment group was the independent variable in the logistic regression; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.64, Regression, Logistic — 2 sided test; Treatment group was the independent variable in the logistic regression
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 48; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.37, Regression, Logistic — 2 sided test; Treatment group was the independent variable in the logistic regression
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 96; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.32, Regression, Logistic; Treatment group was the independent variable in the logistic regression

6. Secondary Outcome: Percentage of Participants With a Sustained Complete Response
Description: The percentage of participants who achieved a sustained complete response, defined as a complete response achieved at Week 48 and Week 96.
  Complete response was defined as meeting all of the following criteria:
  1. Urine protein-to-creatinine ratio (UPCR) < 0.5, based on a 24-hour collection;
  2. Estimated glomerular filtration rate (eGFR) ≥120 ml/min/1.73 m^2 calculated by the CKD-EPI formula or, if < 120 ml/min/1.73 m^2, then > 80% of eGFR at entry; and
  3. Prednisone dose tapered to 10 mg/day and adherence to prednisone dosing provisions.
Time Frame: Week 48, Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants | 26.7 [7.8 to 55.1] | 28.6 [8.4 to 58.1]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 96; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.91, Regression, Logistic — 2 sided test; 2 sided test

7. Secondary Outcome: Percentage of Participants With Treatment Failure by Week 24, Week 48, and Week 96
Description: The percentage of participants who met the criteria for treatment failure, defined by withdrawal from the protocol treatment regimen due to worsening nephritis, infection, or study medication toxicity.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 0 to Week 24 | 18.2 [5.2 to 40.3] | 14.3 [3.1 to 36.3]
  Week 0 to Week 48 | 45.5 [24.4 to 67.8] | 28.6 [11.3 to 52.2]
  Week 0 to Week 96 | 63.6 [40.7 to 82.8] | 47.6 [25.7 to 70.2]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 24; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = .73, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 48; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.26, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 96; Test type: Superiority — Treatment group was the independent variable in the logistic regression; p = 0.29, Regression, Logistic — 2 sided test; 2 sided test

8. Secondary Outcome: Count of Participants: Frequency of Non-renal Flares by Week 24
Description: Count of participants who experienced non-renal flares, defined as any new "A" finding in a non-renal organ system in the British Isles Lupus Assessment Group (BILAG) assessment. A BILAG "A" finding represents a significant increase in, or a new manifestation of, disease activity.
Time Frame: Week 24
Population: The modified intent-to-treat population includes all randomized participants who received 1 dose of Solumedrol, 1 dose of rituximab, 1 dose of cyclophosphamide, and, if in the Rituximab/Cyclophosphamide/Belimumab (RCB) arm, 1 dose of belimumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
Participants
  0 Non-renal flares | 21 | 20
  1 Non-renal flare | 1 | 0
  2 Non-renal flares | 0 | 1
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 24; Test type: Superiority — 2 sided test; p > 0.99, Fisher Exact — 2 sided test; 2 sided test

9. Secondary Outcome: Count of Participants: Frequency of Non-renal Flares by Week 48
Description: as for outcome 8
Time Frame: Week 48
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
Participants
  0 Non-renal flares | 20 | 20
  1 Non-renal flares | 2 | 0
  2 Non-renal flare | 0 | 1
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Week 0 to Week 48; Test type: Superiority — 2 sided test; p = 0.49, Fisher Exact — 2 sided test; 2 sided test

10. Secondary Outcome: Count of Participants: Frequency of Non-renal Flares by Week 96
Description: as for outcome 8
Time Frame: Week 96
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
Participants
  0 Non-renal flares | 18 | 19
  1 Non-renal flare | 4 | 1
  2 Non-renal flares | 0 | 1

11. Secondary Outcome: Percentage of Participants With an Negative Anti-dsDNA Result at Week 24, Week 48, and Week 96
Description: The percentage of participants who were anti-double stranded DNA (anti-dsDNA) negative, defined as having anti-dsDNA levels <30 IU/mL.
  Anti-dsDNA levels are associated with systemic lupus erythematosus disease activity.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 24: number analyzed (Participants) | 21 | 19
  Week 24 | 14.3 [3.1 to 36.3] | 15.8 [3.4 to 39.6]
  Week 48: number analyzed (Participants) | 20 | 20
  Week 48 | 20.0 [5.7 to 43.7] | 30.0 [11.9 to 54.3]
  Week 96: number analyzed (Participants) | 17 | 18
  Week 96 | 0.0 [0.0 to 19.5] | 27.8 [9.7 to 53.5]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — 2 sided test; p = 0.89, Regression, Logistic — 2 sided test
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 48; p = 0.47, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 96; p = 0.94, Regression, Logistic — 2 sided test; 2 sided test

12. Secondary Outcome: Percentage of Participants Hypocomplementemic for Complement Component C3 at Week 24, Week 48, and Week 96
Description: The percentage of participants who were hypocomplementemic for complement component, C3, defined as a C3 level <90 mg/dL.
  Serum C3 complement is a protein which can be measured in the blood. Low blood levels of C3 are common in those with active lupus.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 24: number analyzed (Participants) | 21 | 20
  Week 24 | 57.1 [34.0 to 78.2] | 30.0 [11.9 to 54.3]
  Week 48: number analyzed (Participants) | 20 | 20
  Week 48 | 55.0 [31.5 to 76.9] | 30.0 [11.9 to 54.3]
  Week 96: number analyzed (Participants) | 18 | 18
  Week 96 | 61.1 [35.8 to 82.7] | 27.8 [9.7 to 53.5]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 24; p = 0.08, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 48; p = 0.11, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 96; p = 0.05, Regression, Logistic — 2 sided test; 2 sided test

13. Secondary Outcome: Percentage of Participants Hypocomplementemic for Complement Component C4 at Week 24, Week 48, and Week 96
Description: The percentage of participants who were hypocomplementemic for complemen component C4, defined as a C4 level <10 mg/dL.
  Serum C4 complement is a protein which can be measured in the blood. Low blood levels of C4 are common in those with active lupus.
Time Frame: Week 24, Week 48 and Week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
percentage of participants
  Week 24: number analyzed (Participants) | 21 | 20
  Week 24 | 19.0 [5.5 to 41.9] | 5.0 [0.1 to 24.9]
  Week 48: number analyzed (Participants) | 20 | 20
  Week 48 | 15.0 [3.2 to 37.9] | 15.0 [3.2 to 37.9]
  Week 96: number analyzed (Participants) | 18 | 18
  Week 96 | 16.7 [3.6 to 41.4] | 11.1 [1.4 to 34.7]
Statistical Analysis 1: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 24; p = .20, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 2: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 48; p > 0.99, Regression, Logistic — 2 sided test; 2 sided test
Statistical Analysis 3: Comparison: Rituximab/Cyclophosphamide (RC) vs Rituximab/Cyclophosphamide/Belimumab (RCB); Treatment group was the independent variable in the logistic regression; Test type: Superiority — Week 96; p = 0.63, Regression, Logistic — 2 sided test; 2 sided test

14. Secondary Outcome: Frequency of Specific Adverse Events of Interest By Event by Week 96
Description: Number of ≥ Grade 2 specific treatment-emergent adverse events (AEs) of interest. Grade 2 or higher AEs were classified according to the listed categories of interest based on the study team's review of the AEs.
  Treatment-emergent AEs are those:
  * with an onset date on or after the first dose of study medication,
  * with onset before first dose but that worsened in severity after first dose, and
  * for which the start of the AE in relation to the start of study medication could not be established.
  The severity of AEs was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, v4.03: June 14, 2010). AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 17.0.
Time Frame: Week 96
Population: The safety population includes all participants who received at least one dose of study treatment.
Measure: Number; unit: Events
Groups:
- Rituximab/Cyclophosphamide (RC); Rituximab/Cyclophosphamide/Belimumab (RCB): The safety population includes all participants who received at least one dose of study treatment.
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
Events
  Any event leading to death | 0 | 0
  ≥Grade 2 leukopenia or thrombocytopenia | 13 | 16
  Premature ovarian failure | 0 | 0
  Malignancy | 0 | 0
  Venous thromboembolic event | 3 | 0

15. Secondary Outcome: Frequency of Specific Adverse Events of Interest By Participant, By Week 96
Description: Number of participants who experienced ≥Grade 2 specific treatment-emergent adverse events (AEs) of interest. Grade 2 or higher AEs were classified according to the listed categories of interest based on the study team's review of the AEs.
  Treatment-emergent AEs are those:
  * with an onset date on or after the first dose of study medication,
  * with onset before first dose but that worsened in severity after first dose, and
  * for which the start of the AE in relation to the start of study medication could not be established.
  The severity of AEs was classified using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, v4.03: June 14, 2010). AEs were classified by system organ class and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) version 17.0.
Time Frame: Week 96
Population: The safety population includes all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab/Cyclophosphamide (RC) | Rituximab/Cyclophosphamide/Belimumab (RCB)
Number analyzed (Participants) | 22 | 21
Participants
  Any event leading to death | 0 | 0
  ≥Grade 2 leukopenia or thrombocytopenia | 6 | 6
  Premature ovarian failure | 0 | 0
  Malignancy | 0 | 0
  Venous thromboembolic event | 2 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 8 months (96 Weeks)
Groups:
- RC Group on Treatment; RC Group After Treatment Discontinuation: Participants received infusions of Solumedrol 100mg, rituximab 1000mg, and cyclophosphamide 750mg intravenously (IV) at Week 0 and Week 2. Prednisone 40 mg per day was administered for the first 2 weeks, with a guided steroid taper to 10mg per day by Week 12 and continued treatment until Week 96.
- RCB Group on Treatment; RCB Group After Treatment Discontinuation: Participants received infusions of Solumedrol 100mg, rituximab 1000mg, and cyclophosphamide 750mg intravenously (IV) at Week 0 and Week 2. Prednisone 40 mg per day was administered for the first 2 weeks, with a guided steroid taper to 10mg per day by Week 12 and continued treatment until Week 96. In addition, participants received IV belimumab 10mg/kg at Weeks 4, 6, 8, and then every 4 weeks through Week 48 in addition to prednisone.
Arm/Group | RC Group on Treatment | RCB Group on Treatment | RC Group After Treatment Discontinuation | RCB Group After Treatment Discontinuation
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 6/22 | 4/21 | 8/22 | 1/21
Other Adverse Events (participants affected / at risk) | 22/22 | 21/21 | 11/22 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC Group on Treatment (N=22) | RCB Group on Treatment (N=21) | RC Group After Treatment Discontinuation (N=22) | RCB Group After Treatment Discontinuation (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC Group on Treatment (N=22) | RCB Group on Treatment (N=21) | RC Group After Treatment Discontinuation (N=22) | RCB Group After Treatment Discontinuation (N=21)
Anaemia (Blood and lymphatic system disorders) | 10 (17) | 13 (20) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 5 (10) | 6 (15) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 17 (33) | 11 (19) | 9 (11) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 5 (8) | 2 (2) | 0 (0)
Cushingoid (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 9 (12) | 11 (18) | 4 (5) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (6) | 1 (4) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (7) | 1 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 6 (9) | 8 (11) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (15) | 8 (10) | 2 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 4 (4) | 6 (6) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 7 (7) | 6 (8) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT02260934/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02260934/SAP_001.pdf